CLINICAL TRIAL: NCT00989092
Title: A Randomized, Open-label, Comparative Study to Estimate the Effect of Darbepoetin Alfa on Hospital Days, Economic Outcomes, and Health-related Quality of Life in Subjects With Nonmyeloid Malignancies and Anemia of Cancer
Brief Title: Darbepoetin Alfa and Anemia of Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment and change in product development strategy
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20000219
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Anemia; Anemia of Cancer; Cancer; Carcinoma; Neoplasms; Non-Myeloid Malignancies
Keywords: anemia of cancer; darbepoetin alfa; Aranesp
MeSH Terms: conditions — Anemia; Neoplasms; Carcinoma | interventions — Darbepoetin alfa

ARMS (2):
- Observational Group (Other): Participants in the observation group were evaluated once every 2 weeks for the first 12 weeks (test period). No darbepoetin alfa was administered to the observation group during this period. Darbepoetin alfa could be initiated at a dose of 3.0 μg/kg once every 2 weeks beginning with the first visit after the test period at which the participants hemoglobin concentration was less than or equal to 11.0 g/dL. The dose of darbepoetin alfa could be increased to 5.0 μg/kg once every 2 weeks after 6 weeks of darbepoetin alfa treatment in participants with a hemoglobin change from baseline of less than 1.0 g/dL.
  Interventions: Biological: darbepoetin alfa
- 21 week treatment group (Active Comparator): Participants in the treatment group received darbepoetin alfa subcutaneously (SC) at a dose of 3.0 μg/kg once every 2 weeks for 21 weeks. The dose of darbepoetin alfa could be increased at week 7 (to 5.0 μg/kg once every 2 weeks) or at week 13 (to 9.0 μg/kg once every 2 weeks) in participants with a hemoglobin change from baseline of less than 1.0 g/dL who dose escalated at week 7.
  Interventions: Biological: darbepoetin alfa

INTERVENTIONS:
Biological: darbepoetin alfa — Administered subcutaneously.
  Other Names: Aranesp®

SUMMARY:
This phase 2, multicenter, randomized, open-label, comparative study was designed to determine the effect of darbepoetin alfa on hospital days, economic outcomes, and health related quality of life (HRQOL) in anemic patients with nonmyeloid malignancies who were not receiving chemotherapy. Participants were randomly assigned in a 4:1 allocation ratio to receive either 21 weeks of darbepoetin alfa treatment (treatment group) or 12 weeks of observation followed by up to 9 weeks of darbepoetin alfa treatment (observation group).

ELIGIBILITY:
Inclusion Criteria:

* nonmyeloid malignancies (including lymphocytic leukemias)
* anemia (hemoglobin concentration less than or equal to 11.0 g/dL) due to cancer and/or previous chemotherapy or radiotherapy
* Eastern Cooperative Oncology Group performance status of 0 to 2
* adequate liver and renal functions
* 18 years or older

Exclusion Criteria:

* history of recombinant human erythropoietin therapy, cytotoxic chemotherapy, or more than 30 Gy radiotherapy to the whole pelvis within 4 weeks before screening
* acute myelogenous leukemia, chronic myelogenous leukemia, or myelodysplastic syndrome
* known hematologic disorders that could cause anemia
* inflammatory or cardiac disorders
* previous positive antibody response to any erythropoietic agent
* history of pure red cell aplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2002-05; Primary Completion 2004-01 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Charu V, Belani CP, Gill AN, Bhatt M, Tomita D, Rossi G, Ben-Jacob A. Efficacy and safety of every-2-week darbepoetin alfa in patients with anemia of cancer: a controlled, randomized, open-label phase II trial. Oncologist. 2007 Jun;12(6):727-37. doi: 10.1634/theoncologist.12-6-727. PMID 17602062
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Randomized: 24-Jun-2002 Last Patient Randomized: 08-Aug-2003
Groups:
- Darbepoetin Alfa 3 μg/kg: Participants in the treatment group received darbepoetin alfa subcutaneously (SC) at a dose of 3.0 μg/kg once every 2 weeks for 21 weeks. The dose of darbepoetin alfa could be increased at Week 7 (to 5.0 μg/kg once every 2 weeks) or at Week 13 (to 9.0 μg/kg once every 2 weeks) in participants with a hemoglobin change from baseline of less than 1.0 g/dL who dose escalated at Week 7.
- Observation: Participants in the observation group were evaluated once every 2 weeks for the first 12 weeks (test period). No darbepoetin alfa was administered during this period. Darbepoetin alfa could be initiated at a dose of 3.0 μg/kg once every 2 weeks beginning with the first visit after the test period at which the participant's hemoglobin concentration was less than or equal to 11.0 g/dL. The dose of darbepoetin alfa could be increased to 5.0 μg/kg once every 2 weeks after 6 weeks of darbepoetin alfa treatment in participants with a hemoglobin change from baseline of less than 1.0 g/dL.
Period: Overall Study
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Started | 228 | 59
Treated With Darbepoetin Alfa | 226 | 33
Completed | 138 | 31
Not Completed | 90 | 28
Not completed — Physician Decision | 9 | 6
Not completed — Adverse Event | 20 | 1
Not completed — Chemotherapy initiated | 12 | 4
Not completed — Withdrawal by Subject | 17 | 9
Not completed — Death | 14 | 2
Not completed — Ineligibility determined | 3 | 3
Not completed — Lost to Follow-up | 6 | 2
Not completed — Other | 3 | 1
Not completed — Protocol deviation | 2 | 0
Not completed — Erythropoietin therapy initiated | 2 | 0
Not completed — Did not receive study drug | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation | Total
Number analyzed (Participants) | 226 | 59 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] — Demographic data are provided for the Efficacy Analysis Set (all patients who were randomized to the observation group or patients who were randomized to the treatment group and received at least 1 dose of investigational product).
  Years | 71.7 (10.4) | 67.2 (12.5) | 70.8 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 36 | 167
  Male | 95 | 23 | 118
Race/Ethnicity, Customized [Number; unit: Participant]
  White | 188 | 46 | 234
  Black | 28 | 12 | 40
  Asian | 5 | 1 | 6
  Other | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Hospitalized During the Test Period
Description: Number of participants hospitalized during Weeks 1-12 as self-reported in the Health Care Utilization portion of the Subject Outcome Questionaire.
Time Frame: Weeks 1- 12
Population: Includes all randomized patients in the darbepoetin alfa arm who received at least 1 dose of study drug or all randomized patients in the observation arm. Patients also needed to have completed the baseline and at least 1 post-baseline subject outcome questionaire.
Measure: Number; unit: Participants
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 215 | 45
Participants | 23 | 6

2. Secondary Outcome: Total Hospital Costs During the Test Period
Description: The hospital bill database was used to determine the mean total hospital cost per participant during the test period. Participants who were not hospitalized had a cost of $0 imputed.
Time Frame: Weeks 1-12
Population: Includes all randomized patients in the darbepoetin alfa arm who received at least 1 dose of study drug or all randomized patients in the observation arm, and were included in the hospital bill database. Participants who were not hospitalized had a cost of $0 imputed.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 198 | 40
dollars | 1474.58 (5528.61) | 487.31 (1821.43)

3. Secondary Outcome: Change in Functional Assessment of Cancer Therapy (FACT)-Fatigue Score at Week 13
Description: The FACT-Fatigue scale comprises 13 questions evaluating the impact of anemia on cancer patients with various tumor types receiving chemotherapy. Fatigue scores range from 0 to 52, with a higher score indicating less fatigue.
Time Frame: Baseline (Week 1) and Week 13
Population: Includes all randomized patients in the darbepoetin alfa arm who received at least 1 dose of study drug or all randomized patients in the observation arm. Participants also needed to have completed the baseline and at least 1 post-baseline FACT-Fatigue questionaire. Last Value Carried Forward (LVCF) imputation used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 215 | 45
units on a scale | 6.0 (12.0) | 2.2 (7.6)

4. Secondary Outcome: Hemoglobin Response During the Test Period
Description: The number of participants achieving a hemoglobin response, defined as an increase in hemoglobin from baseline of ≥ 2.0 g/dL in the absence of red blood cell (RBC) transfusions during the preceding 28 days.
Time Frame: Weeks 1-12
Population: Includes all randomized patients in the darbepoetin alfa arm who received at least 1 dose of study drug or all randomized patients in the observation arm. Patients also needed to have a baseline hemoglobin that was not affected by a red blood cell transfusion.
Measure: Number; unit: Participants
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 220 | 55
Participants | 128 | 4

5. Secondary Outcome: Hematopoietic Response During the Test Period
Description: The number of participants achieving a hematopoietic response, defined as an increase in hemoglobin from baseline of ≥ 2.0 g/dL or a concentration ≥ 12.0 g/dL both in the absence of red blood cell (RBC) transfusions during the preceding 28 days.
Time Frame: Weeks 1-12
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 220 | 55
Participants | 145 | 10

6. Secondary Outcome: Change From Baseline in Hemoglobin Level
Description: The difference between hemoglobin concentrations after 12 weeks of treatment and the Baseline hemoglobin concentration value (Study Day 1 sample prior to first dose of darbepoetin alfa).
Time Frame: Baseline (Week 1) and Week 13
Population: Includes all randomized patients in the darbepoetin alfa arm who received at least 1 dose of study drug or all randomized patients in the observation arm. Patients also needed to have a baseline hemoglobin that was not affected by a red blood cell transfusion. LVCF imputation was used.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 220 | 55
g/dL | 2.1 (1.9) | 0.1 (0.8)

7. Secondary Outcome: Number of Participants With Red Blood Cell (RBC) Transfusions During the Test Period
Description: Number of participants with at least one RBC transfusion during Weeks 1 to 12.
Time Frame: Weeks 1-12
Population: Includes all randomized patients in the darbepoetin alfa arm who received at least 1 dose of study drug or all randomized patients in the observation arm with available data.
Measure: Number; unit: Participants
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 226 | 59
Participants | 25 | 11

8. Primary Outcome: Days of Hospitalization During the Test Period
Description: Number of days hospitalized during Weeks 1-12 as self-reported in the Health Care Utilization portion of the Subject Outcome Questionaire; participants who were not hospitalized had a value of 0 days.
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 212 | 44
days | 0.5 (2.2) | 0.5 (1.7)

9. Primary Outcome: Number of Hospitalizations During the Test Period
Description: Number of times participants were hospitalized as self-reported in the Health Care Utilization portion of the Subject Outcome Questionaire during Weeks 1-12
Time Frame: Weeks 1-12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 215 | 45
hospitalizations | 0.1 (0.5) | 0.2 (0.4)

10. Secondary Outcome: Number of Units of Red Blood Cells Transfused During the Test Period
Description: The average number of standard units of red blood cells transfused during Weeks 1 to 12.
Time Frame: Weeks 1-12
Population: Includes all randomized patients in the darbepoetin alfa arm who received at least 1 dose of study drug or all randomized patients in the observation arm.
Measure: Mean (Standard Deviation); unit: units of red blood cells
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 226 | 59
units of red blood cells | 0.4 (1.4) | 0.9 (2.4)

11. Secondary Outcome: Number of Days of Red Blood Cell Transfusions During the Test Period
Description: The number of days when at least one red blood cell transfusion was administered during Weeks 1 to 12.
Time Frame: Weeks 1-12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 226 | 59
days | 0.2 (0.6) | 0.4 (1.0)

12. Secondary Outcome: Number of Participants With Red Blood Cell (RBC) Transfusions During Weeks 5-12
Description: The number of participants with at least one RBC transfusion during weeks 5 to 12.
Time Frame: Weeks 5-12
Population: Includes all randomized patients in the darbepoetin alfa arm who received at least 1 dose of study drug or all randomized patients in the observation arm, and who were on-study as of the beginning of Week 5 (Study Day 29).
Measure: Number; unit: Participants
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 215 | 47
Participants | 16 | 10

13. Secondary Outcome: Number of Units of Red Blood Cells Transfused During Weeks 5-12
Description: The number of standard units of RBCs transfused during Weeks 5 to 12.
Time Frame: Weeks 5-12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units of red blood cells
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 215 | 47
units of red blood cells | 0.2 (1.0) | 0.8 (1.8)

14. Secondary Outcome: Number of Days of Red Blood Cell Transfusions During Weeks 5-12
Description: The number of days when at least one RBC transfusion was administered during Weeks 5 to 12.
Time Frame: Weeks 5-12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Darbepoetin Alfa 3 μg/kg | Observation
Number analyzed (Participants) | 215 | 47
days | 0.1 (0.5) | 0.4 (0.8)

ADVERSE EVENTS:
Time Frame: First dose through End of Study or 30 days after last dose, up to 25 weeks.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Groups:
- Treatment Arm: Participants in the treatment group received darbepoetin alfa subcutaneously (SC) at a dose of 3.0 μg/kg once every 2 weeks for 21 weeks. The dose of darbepoetin alfa could be increased at week 7 (to 5.0 μg/kg once every 2 weeks) or at week 13 (to 9.0 μg/kg once every 2 weeks) in participants with a hemoglobin change from baseline of less than 1.0 g/dL who dose escalated at week 7.
- Observation Arm Treated: Participants in the observation group who received darbepoetin alfa, initiated at a dose of 3.0 μg/kg once every 2 weeks beginning with the first visit after the test period at which the participants hemoglobin concentration was less than or equal to 11.0 g/dL. The dose of darbepoetin alfa could be increased to 5.0 μg/kg once every 2 weeks after 6 weeks of darbepoetin alfa treatment in participants with a hemoglobin change from baseline of less than 1.0 g/dL. Adverse events for participants in this group could have been reported at any time during the study; and therefore, may have occurred before darbepoetin alfa administration.
- Observation Arm Not Treated: Participants in the observation group who did not receive any darbepoetin alfa treatment.
Arm/Group | Treatment Arm | Observation Arm Treated | Observation Arm Not Treated
Serious Adverse Events (participants affected / at risk) | 65/226 | 4/33 | 4/26
Other Adverse Events (participants affected / at risk) | 99/226 | 21/33 | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=226) | Observation Arm Treated (N=33) | Observation Arm Not Treated (N=26)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 0
Asthenia (General disorders) | 4 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Gastrostomy tube insertion (Surgical and medical procedures) | 1 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=226) | Observation Arm Treated (N=33) | Observation Arm Not Treated (N=26)
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 13 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 16 | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 0
Asthenia (General disorders) | 22 | 2 | 2
Fatigue (General disorders) | 42 | 6 | 3
Oedema peripheral (General disorders) | 20 | 1 | 1
Pain (General disorders) | 9 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
Dizziness (Nervous system disorders) | 12 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 6 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hot flush (Vascular disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.